CLINICAL TRIAL: NCT00259844
Title: A Phase 2 Study Immunologically Evaluating 5T4-MVA (TroVax) in Patients Undergoing Surgical Resection of Colorectal Liver Metastases
Brief Title: Effect of TroVax in Patients Having Colorectal Cancer With Liver Metastases Removed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: Oxford BioMedica (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH2/048
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2006-07-18 (Estimated); Status verified 2005-11

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal; Liver Metastases; Vaccine; Colorectal Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — TroVax

INTERVENTIONS:
Biological: TroVax

SUMMARY:
This study will test the safety and efficacy of TroVax in patients undergoing surgical resection of colorectal cancer with liver metastases.

TroVax potentially works by encouraging the immune system to react against the 5T4 protein on the surface of bowel cancer cells. The immune system is then able to recognise 5T4 and kill cells that carry it. The hope is that if tumour cells started to grow again after the main tumour has been surgically removed, the immune system would be able to find and destroy them.

DETAILED DESCRIPTION:
Treatment of metastatic colorectal cancer depends on the site of disease. The prognosis for patients is poor although cure can be obtained if disease is localised and operable. Patients with metastatic disease confined to the liver may achieve a cure rate of between 20% and 60% if these metastases are resited, but there is a risk that micrometastatic disease will persist post-operatively.

TroVax consists of a highly attenuated vaccinia virus (modified vaccinia Ankara) containing the human tumour associated antigen ST4.

The human oncofetal antigen 5T4 a surface glycoprotein expressed by placental tissue, but also by a wide range of human carcinomas including most colorectal and renal carcinomas. 5T4 exhibits only low level expression in normal tissue and is thus a suitable target for immune therapy of cancer.

This study will evaluate for the first time in man the immunological effects of the TroVax vaccine locally within a target tumour and in peripheral blood. Tolerability of the vaccine will also be assessed.

Patients receive 2 intramuscular injections of TroVax at a 2 week interval followed by surgery 10 days later. Two further vaccinations are given at 4 and 8 weeks after surgery. Patients who show a response to the first four vaccinations are given 2 additional vaccinations 20 and 28 weeks post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal adenocarcinoma with metastases confined only to the liver, histologically proven and considered suitable for treatment by surgical resection.
* World Health Organisation (WHO) performance status of 0 or 1
* All toxic manifestations of previous treatment must have resolved. Exceptions to this are alopecia or certain Grade 1 toxicities which in the opinion of the Investigator and Cancer Research UK should not exclude the patient.

Exclusion Criteria:

* Radiotherapy, endocrine therapy, immunotherapy, systemic steroids, or chemotherapy during the previous four weeks (six weeks for nitrosoureas and Mitomycin-C) prior to treatment or during the course of the trial.
* Patients who are high medical risks because of non-malignant systemic disease, including those with active uncontrolled infection.
* Concurrent serious infections within the 28 days prior to entry to the trial
* Current malignancies at other sites, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.
* Patients known to be serologically positive for Hepatitis B, C or HIV
* History of allergy to vaccinations or egg proteins.
* Inflammatory bowel disease
* History of autoimmune disease
* Clinical evidence of cerebral metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-06; Study Completion 2006-12

PRIMARY OUTCOMES:
To characterise and quantify the immune response to the oncofetal antigen 5T4 locally in peripheral blood, modified by vaccination with TroVax before resection of colorectal adenocarcinoma liver metastases.
To evaluate the safety, toxicity and tolerability of the TroVax vaccine in this setting.

SECONDARY OUTCOMES:
To characterise and quantify the immune response to the oncofetal antigen 5T4 locally in tumour.
To review any further effect on immunity by TroVax vaccinations following surgery.
To monitor and collect data on clinical outcomes (time to progression/relapse/death).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hawkins, MD, Prof, Principal Investigator — The Christie NHS Foundation Trust